CLINICAL TRIAL: NCT05085769
Title: Potential Associations Between Alterations in Gut Microbiome and Obesity-related Traits After the Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Ozdemir, Research Assistant, Hacettepe University
Other Study IDs: GO14/533
Record Dates: First submitted 2021-09-07; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Bariatric Surgery
Keywords: obesity; bariatric surgery; gut microbiome; diet
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study group: 15 patients who had bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Control group-1: 8 morbidly obese participants who did not have bariatric surgery
- Control group-2: 11 participants who were non-obese

INTERVENTIONS:
Procedure: Bariatric surgery — A procedure for morbidly obese patients whose body mass index (BMI) is higher than 40 kg/m2 or 35 kg/m2 and having comorbidities of obesity.
  Groups: Study group

SUMMARY:
This study aimed to examine the effects of obesity and bariatric surgery on gut microbiota in a Turkish population, and to contribute to the literature by bringing multi-dimensional parameters including dietary intake, metabolic and inflammatory markers. This case-control study was conducted between June 2015 and August 2019. All participants were followed during the six-month period. Face-to-face interviews and physical examinations were held, and blood and fecal samples were collected at the baseline (M0) and at the end of 3 (M3) and 6 months (M6). Dietary intakes of subjects were assessed using 24-h dietary recall method in each interview and a detailed quantitative food frequency questionnaire that involved 85 food items. Subjects were recruited to the study as three groups: 15 patients who had bariatric surgery as study group, 8 morbidly obese participants who did not have bariatric surgery as control group-1 and 11 participants who were non-obese (lean (n=5) and pre-obese (n=6)) as control group-2. All subjects in the study group had sleeve gastrectomy. Subjects in control groups were selected as age and gender matched with the participants in the study group. Individuals were excluded if (a) they were under 19 or above 65 years old, (b) they had an acute or chronic inflammatory disease, (c) they were diagnosed with infectious diseases, cancer or alcohol addiction, (d) they used antibiotics in last 3 months before the screening.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese participants for study and control group-1
* non-obese participants for control group-2

Exclusion Criteria:

* they were under 19 or above 65 years old,
* they had an acute or chronic inflammatory disease,
* they were diagnosed with infectious diseases, cancer or alcohol addiction,
* they used antibiotics in last 3 months before the screening.

Ages: 26 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects were recruited to the study as three groups: 15 patients who had bariatric surgery as study group, 8 morbidly obese participants who did not have bariatric surgery as control group-1 and 11 participants who were non-obese (lean (n=5) and pre-obese (n=6)) as control group-2.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbial profiles of participants | 6 months
  Changes in bacterial phyla and sub-phylum levels
Changes in gut bacterial biodiversity of participants | 6 months
  Changes in gut bacterial alpha and beta biodiversity of participants

SECONDARY OUTCOMES:
Changes in dietary energy and nutrient intakes | 6 months
  Changes in dietary energy in calories, macro-, micronutrient intakes in grams
Changes in food intakes | 6 months
  Changes in certain food groups in grams

OTHER OUTCOMES:
Changes in body weight | 6 months
  Changes in body weight in kilograms
Changes in body mass index | 6 months
  Changes in body mass index in kg/m^2
Changes in body fat and fat free mass | 6 months
  Changes in fat mass and fat free mass in kilograms
Changes in waist circumferences | 6 months
  Changes in waist circumferences in centimeters
Changes in serum glucose levels | 6 months
  Changes in serum glucose in mg/dL
Changes in lipid related biochemical parameters | 6 months
  Changes in triglyceride, total cholesterol, LDL cholesterol, HDL cholesterol levels in mg/dL
Changes in liver function tests | 6 months
  Changes in ALT and AST levels in U/L
Changes in serum IL-6 and TNF-alpha levels | 6 months
  Changes in serum IL-6 and TNF-alpha levels in ng/mL
Changes in serum hs-CRP levels | 6 months
  Changes in serum hs-CRP in mg/L

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir A, Sarzhanov F, Dogruman-Al F, Gundogdu A, Nalbantoglu U, Yozgat A, Yildiz BD, Buyuktuncer Z. Exploring the complex interplay of Blastocystis, morbid obesity, and bariatric surgery on gut microbial dynamics. Microb Pathog. 2025 Mar;200:107306. doi: 10.1016/j.micpath.2025.107306. Epub 2025 Jan 15. PMID 39824262